CLINICAL TRIAL: NCT05518240
Title: Comparison of Solitaire to Embotrap to Treat Large Vessel Occlusion in Acute Ischemic Stroke (SOLTRAP Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: WellStar Health System (Other)
Responsible Party: Principal Investigator, Benjamin Zussman, MD, Comparison of Solitaire to Embotrap to treat Large Vessel Occlusion in Acute Ischemic stroke (SOLTRAP Study), WellStar Health System
Other Study IDs: Sol9058
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acute ischemic stroke (AIS): Patients who experienced acute ischemic stroke (AIS), eligible for restoration of blood flow using a Solitaire or Embotrap device to remove thrombus from the neurovasculature
  Interventions: Device: Stent Retrievers; Device: Stent Retriever

INTERVENTIONS:
Device: Stent Retrievers — Procedure: Embotrap device
Device: Stent Retriever — Procedure: Solitaire device

SUMMARY:
The primary aim of this study is to assess if there is a difference in first pass reperfusion between the two devices. This is a randomized prospective study to assess if there is a difference in first pass reperfusion at two centers with large mechanical thrombectomy volumes. Data will also be collected on time-to treatment, outcomes and hemorrhagic complications.

DETAILED DESCRIPTION:
The SOLTRAP Study is an investigator initiated two hospital study designed to assess the procedural success and clinical outcomes associated with mechanical thrombectomy using the Medtronic Solitaire Device and the Cerenovous Embotrap device. Both devices are FDA approved for this indication of removal of a thrombus for patients suffering from stroke secondary to a large vessel occlusion.

Data collected will include device used during the procedure, mechanical thrombectomy techniques, time from onset to imaging, imaging to puncture, and overall time from onset to reperfusion as well as quality of life at 90 days post stroke.

The study will enroll up to 418 subjects and will be conducted at Wellstar North Fulton Hospital and Wellstar Kennestone Hospital. The devices will have regulatory authorization to be on the market in the geographic location of both sites.

The duration of the Registry protocol is approximately 24 months

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who experienced acute ischemic stroke (AIS), eligible for restoration of blood flow using a Solitaire or Embotrap device to remove thrombus from the neurovasculature
2. Occlusion of intracranial cerebral circulation vessel involving the M1, M2 MCA or ICA-T (Tandem occlusions will be enrolled)
3. Subject or subject's legally authorized representative (LAR) has signed the informed consent form prior to or within 72 hours post-procedure
4. Subject is willing to comply with the protocol follow-up requirements
5. The intended technique and treated technique must be one of the following techniques for the first thrombectomy pass in the neurovasculature per Instructions for Use (IFU).

Exclusion Criteria:

1.The subject can participate in another clinical trial if the study does not impact the endpoints defined in this protocol given this is a data collection trial. Patients who are unable to comply wit the 90 day follow up in person or via telephone will be excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who experienced acute ischemic stroke (AIS), eligible for restoration of blood flow using a Solitaire or Embotrap device to remove thrombus from the neurovasculature
Sampling Method: Probability Sample
Enrollment: 418 (Estimated)
Dates: Start 2022-08-24 (Estimated); Primary Completion 2024-08-07 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Severity of Disability | Day 90 (+14)
  assessed by mRS with a good functional outcome defined as mRS of 0-2 for each technique

SECONDARY OUTCOMES:
Excellent functional outcome | Day 90 (+14)
  defined as mRS 0-1 at Day 90

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Wellstar North Fulton Hospital, Roswell, Georgia

IPD SHARING:
Plan to Share IPD: No